CLINICAL TRIAL: NCT00216749
Title: Post Marketing Surveillance of Efficacy and Safety of Cilostazol for the Indication of CSPS
Brief Title: Efficacy and Safety of Cilostazol for the Indication of CSPS
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Clinical Reserch Team Leader, Korea Otsuka Pharmaceutical Co. Ltd
Other Study IDs: Korea Pletaal CSPS PMS
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Cerebral Infarction
Keywords: Cerebral Infarction Prevention; Cilostazol
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cilostazol: Cilostazol Treatment Patients who were in stable states after the occurrence of cerebral infarction (except cardiogenic cerebral embolism)

SUMMARY:
This is a multicenter, open-label, prospective study of cilostazol use for prevention of recurrence in patients with cerebral infarction.

DETAILED DESCRIPTION:
This is a multicenter, open-label, prospective study of cilostazol use to prevention of recurrence in patients with cerebral infarction.

Qualified patients will be treated with cilostazol by physician's assessment. This study will be continued for 4 years. More than 600 patients for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an experience of cerebral infarction and having a purpose for prevention of recurrence of cerebral infarction.
* Age: more than 18 years of age

Exclusion Criteria:

* Unqualified patients judged by study investigator(s)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in restabilization status after cerebral infarction (excluding cardiogenic cerebral embolism)
Sampling Method: Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
1)Efficacy:Recurrence of cerebral infarction 2)Safety:Adverse Event | 3M

CONTACTS AND LOCATIONS:
Overall Officials: Bo Youn Seo, Study Director — Korea Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Asan Medical Center, Seoul, South Korea